CLINICAL TRIAL: NCT07394478
Title: Study of the Association Between Sacroiliitis/Axial Spondylarthritis and Giant Cell Arteritis/ Polymyalgia Rheumatica: A Case-control Observational Study
Brief Title: Study of the Association Between Sacroiliitis/Axial Spondylarthritis and Giant Cell Arteritis/ Polymyalgia Rheumatica
Acronym: SAGE PPR
Status: Not yet recruiting | Type: Observational
Sponsor: Hôpital NOVO (Other)
Collaborators: GEFA (Unknown); CRI (Unknown)
Responsible Party: Sponsor
Other Study IDs: CHRD 1625
Record Dates: First submitted 2026-01-27; First posted 2026-02-06 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Giant Cell Arteritis (GCA); Spondylarthritis; Polymyalgia Rheumatica
Keywords: Giant Cell Arteritis (GCA); Spondylarthritis; Polymyalgia rheumatica
MeSH Terms: conditions — Giant Cell Arteritis; Spondylarthritis; Polymyalgia Rheumatica

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with GCA, spondylarthritis and/or polymyalgia rheumatica: Patients with GCA, spondylarthritis and/or polymyalgia rheumatica
  Interventions: Other: Description of population

INTERVENTIONS:
Other: Description of population — Description of population in the aim of identify demographic or phenotypic factors different between experimental and control populations.

SUMMARY:
The purpose of the study is to recruit as many patients as possible presenting with sacroiliitis or authentic axial spondylarthritis and giant cell arteritis. The investigators will also be interested in the association of spondylarthritis and polymyalgia rheumatica given the continuum between these two pathologies. The aim is to investigate whether there is an association between giant cell arteritis and spondylarthritis or polymyalgia rheumatica and spondylarthritis.

DETAILED DESCRIPTION:
Large vessel vasculitis primarily includes Takayasu's arteritis and Giant Cell Arteritis (GCA). The literature describes associations between spondyloarthritis and large vessel vasculitis, particularly with Takayasu's arteritis. Case reports have highlighted specific features in patients presenting with both conditions, such as an older age at spondyloarthritis diagnosis and higher C-reactive protein (CRP) levels, for example.

However, to date, no cases of axial spondyloarthritis associated with confirmed GCA have been reported in the literature.

The investigators plan to recruit cases (patients with GCA and/or polymyalgia rheumatica [PMR] plus spondyloarthritis) and controls (patients with GCA or PMR alone). The investigators will then analyze their characteristics to investigate a potential association between these diseases.

ELIGIBILITY:
Inclusion Criteria:

* Experimental group: Adult patient with spondylitis associated with GCA or PMR Control group: Adult patient with GCA or PMR

Exclusion Criteria:

* Refusal to participate
* Positive anti CCP

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: - Experimental group: Adult patient with spondylitis associated with GCA or PMR Control group: Adult patient with GCA or PMR
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Description of the population of patients with spondylarthritis associated with giant cell arteritis (GCA) or polymyalgia rheumatica (PMR) versus patients with GCA or PMR alone | At baseline
  Identification of demographic or phenotypic factors different between experimental and control populations.

CONTACTS AND LOCATIONS:
Overall Officials: Omar AL TABAA, Principal Investigator — Hôpital NOVO; Auriane CHADELAT, Principal Investigator — Hôpital NOVO
Locations (2):
- France (2):
  - CRI (Rheumatism and Inflammatory Club), Paris
  - GEFA (French Group for the study of large vessel Arteritis), Toulouse

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] L.A. Healey, Relation of giant cell arteritis to polymyalgia rheumatica, Baillière's Clinical Rheumatology, Volume 5, Issue 3, 1991, Pages 371-378, ISSN 0950-3579
- [Background] Aydeniz A, Akaltun MS, Gur A, Gursoy S. [Coexistence of polymyalgia rheumatica with ankylosing spondylitis: A case report]. Agri. 2018 Jan;30(1):35-37. doi: 10.5505/agri.2016.69672. Turkish. PMID 29450875
- [Background] Corli J, Lemeunier L, le Gouellec N, Flipo RM. Giant cell arteritis occurring during psoriatic arthritis treated by adalimumab. Joint Bone Spine. 2015;82:291-2.
- [Background] 13 Clementz GL, Gold F, Khaiser N, ZolinWD, Jalovec L. Giant cell arteritis associated with pericarditis and pancreatic insufficiency in a patient with psoriatic arthritis. Rheumatol. 1989;16:128-9.
- [Background] 12 Aortitis due to Giant Cell Arteritis and Psoriatic Arthritis: An Uncommon Association M. del Pilar García-Cezón de la Cruz,a Raquel Almodóvar,b,∗Javier García Pérez,c Patricia Fanny Dhimes,d Pedro Zarcob DOI: 10.1016/j.reumae.2016.03.013
- [Background] Elkayam O, Paran D, Yaron M, Caspi D. Polymyalgia rheumatica in patients with ankylosing spondylitis: a report of 5 cases. Clin Exp Rheumatol. 1997;15:411-4.
- [Background] Eshed I, Druyan A, Stern M, Bordavka M, Lidar M. The prevalence of sacroiliitis on abdominal MRI examinations of patients with Takayasu arteritis. Acta Radiol. 2022 Mar;63(3):387-392. doi: 10.1177/0284185121996270. Epub 2021 Apr 11. PMID 33843285
- [Background] 8. Pawel Mielnik, Anja Myhre Hjelle, Jan Leidulv Nordeide, Coexistence of Takayasu's arteritis and ankylosing spondylitis may not be accidental - Is there a need for a new subgroup in the spondyloarthritis family?, Modern Rheumatology, Volume 28, Issue 2, 4 March 2018, Pages 313-318, https://doi.org/10.1080/14397595.2017.1341592 2018 Mar;28(2):313-318. doi: 10.1080/14397595.2017.1341592. Epub 2017 Jul 18.
- [Background] 7. Abacar, K., Kaymaz-Tahra, S., Bayındır, Ö. et al. Frequency and the effects of spondyloarthritis-spectrum disorders on the clinical course and management of Takayasu arteritis: an observational retrospective study. Clin Rheumatol 43, 1571-1578 (2024). https://doi.org/10.1007/s10067-024-06939-y
- [Background] Riviere E, Arnaud L, Ebbo M, Allanore Y, Claudepierre P, Dernis E, Ziza JM, Miceli-Richard C, Philippe P, Richez C, Soubrier M, Belkhir R, Seror R, Mariette X, Pavy S; Club Rhumatismes et Inflammations. Takayasu Arteritis and Spondyloarthritis: Coincidence or Association? A Study of 14 Cases. J Rheumatol. 2017 Jul;44(7):1011-1017. doi: 10.3899/jrheum.160762. Epub 2017 Apr 15. PMID 28412700
- [Background] Gan FY, Fei YY, Li MT, Wang Q, Xu D, Hou Y, Zeng XF, Zhang FC. The characteristics of patients having ankylosing spondylitis associated with Takayasu's arteritis. Clin Rheumatol. 2014 Mar;33(3):355-8. doi: 10.1007/s10067-013-2444-7. Epub 2013 Dec 6. PMID 24310108
- [Background] 4. Güzel Esen S, Armagan B, Atas N, Ucar M, Varan Ö, Erden A et al (2019) Increased incidence of spondyloarthropathies in patients with Takayasu arteritis: a systematic clinical survey. Joint Bone Spine 86(4):497-501. https://doi.org/10.1016/j.jbspin.2019. 01.020
- [Background] 3. Kwon OC, Lee SW, Park YB, Oh JS, Lee SH, Hong S et al (2018) Extravascular manifestations of Takayasu arteritis: focusing on the features shared with spondyloarthritis. Arthritis Res Ther. 20(1):142. https://doi.org/10.1186/s13075-018-1643-7
- [Background] 2. Momeni M, Taylor N and Tehrani M. Cardiopulmonary manifestations of ankylosing spondylitis. Int J Rheumatol 2011; 2011: 728471
- [Background] 1. Ozkan Y. Cardiac involvement in ankylosing spondylitis. J Clin Med Res 2016; 8: 427-430